CLINICAL TRIAL: NCT06218940
Title: A Phase 1, Open-label, Multicenter Study to Evaluate Safety, Tolerability, PK, and Efficacy of Intravenous Administration of HY1272 in Patients With Late Phase Solid Tumors or EGFRm+NSCLC
Brief Title: HY1272 in Patients With Locally Advanced or Metastatic Solid Tumors or Locally Advanced or Metastatic EGFRm+ NSCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY1271-12-01
Record Dates: First submitted 2024-01-05; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HY1272 (Experimental): HY1272 IV weekly
  Interventions: Drug: HY1272

INTERVENTIONS:
Drug: HY1272 — Each patient will receive HY1272 weely or HY1272 weely+Oshitinib 80mg P.O. daily

SUMMARY:
This is a Phase 1, open-label, multicenter, dose escalation study of HY1272 (administered via IV) evaluating both Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) in patients diagnosed with locally advanced or metastatic solid tumors (monotherapy) or locally advanced or metastatic EGFRm+ NSCLC (combination therapy). The study is designed to evaluate safety, tolerability, PK, and anti-tumor activity of HY1272 administered once weekly. Patients in the monotherapy portion of this study will receive only HY1272. Patients in the combination therapy portion of this study will receive osimertinib administered once daily (QD) with HY1272.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study-specific procedures, sampling, and analyses. If a patient declines to participate in any voluntary exploratory research and/or genetic component of the study, there will be no penalty or loss of benefit to the patient, and they will not be excluded from other aspects of the study.
2. At least 18 years of age.
3. Histological or cytological confirmed diagnosis of locally advanced or metastatic solid tumor(s)
4. All patients must have documented EGFRm+, prior to enrolling in the combination therapy cohorts of this study.
5. All patients must be eligible for treatment with osimertinib prior to enrolling in the combination therapy portion of this study.
6. World Health Organization (WHO) performance status equal to 0-2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
7. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study Screening period, and that can be accurately measured at Baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), which is suitable for accurately repeated measurements.

Exclusion Criteria:

1. Treatment with any of the following:

   1. An EGFR TKI (e.g., erlotinib, gefitinib, or osimertinib) within 8 days or approximately 5× the half-life of the specific drug, whichever is longer, of the first dose of study treatment. (If sufficient wash-out time has not occurred due to scheduling or PK properties, an alternative appropriate wash-out time based on known duration and time to reversibility of drug-related adverse events must be agreed upon by the Sponsors and the Investigator).
   2. Any cytotoxic chemotherapy, investigational agents, or anticancer drugs used for a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
   3. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
   4. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment.
2. Previously untreated NSCLC patients. To be enrolled into the combination therapy cohorts, patients must be eligible to be treated with osimertinib.
3. Any unresolved toxicities from prior therapy >Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or greater at the time of starting study treatment, with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy.
4. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study treatment.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diathesis, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus [HIV]). Screening for chronic conditions is not required.
6. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) >470 msec obtained from 3 electrocardiograms (ECGs), using the Screening clinic ECG machine and Fridericia's formula for QT interval correction.
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives, or any concomitant medication known to prolong the QT interval.
7. Past medical history of EGFR TKI-related interstitial lung disease, except other interstitial lung disease which is not clinically active within last 6 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Evalute safety, tolerability of HY1272 in patients from day 1 to end of study. | baseline to study end （24 months as planned）
  Incidence and severity of various adverse events, including physical examination, blood routine, blood biochemistry, urine flow sediment test, coagulation function, vital signs (pulse, respiration, blood pressure, body temperature), electrocardiogram, etc
Evalute PK of HY1272 in patients from week 1 to week 3. | Week 1 to week 3.
  Evaluate changes of Pharmacokinetics (PK) evaluation mainly Cmax from Week 1 to Week 3.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Chen, Study Director — Sponsor GmbH